CLINICAL TRIAL: NCT01960179
Title: An Open-label, Multicenter 24-Week And 52-Week Study Assessing The Safety And Tolerability Of Lixisenatide In Monotherapy In Patients With Type 2 Diabetes
Brief Title: Safety And Tolerability Of Lixisenatide In Monotherapy In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFY13476; U1111-1134-2695 (Other: UTN)
Record Dates: First submitted 2013-09-27; First posted 2013-10-10 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lixisenatide (Experimental): lixisenatide monotherapy by group (Group 1: 52-week treatment; Group 2: 24-week treatment)
  Interventions: Drug: lixisenatide AVE0010

INTERVENTIONS:
Drug: lixisenatide AVE0010 — Pharmaceutical form:solution Route of administration: Subcutaneous injection

SUMMARY:
Primary Objective:

To assess the overall safety of lixisenatide once daily treatment in monotherapy over 24 and 52 weeks in patients with type 2 diabetes in Japan

Secondary Objective:

To assess the effects of lixisenatide once daily treatment in monotherapy over 24 and 52 weeks on:

* HbA1c (Glycated hemoglobin A1c) reduction;
* Fasting plasma glucose;
* Body weight.

DETAILED DESCRIPTION:
* Group 1: 60 weeks ± 11 days
* Group 2: 32 weeks ± 7 days

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes mellitus diagnosed for at least 2 months.
* Not treated with anti-diabetic drug or treated with a stable dose of 1 oral anti-diabetic drug (OAD) for at least 3 months prior to screening visit. Previous OAD (if any) have to be stopped at Visit 1.1 to be washed out during the run-in period at least for 6 weeks;
* Signed written informed consent.

Exclusion criteria:

* At screening
* age <20 years;
* HbA1c <7% or >9.5% (for patients on OAD <6.5% or >8.5%);
* fasting plasma glucose >250 mg/dL (>13.9 mmol/L);
* Use of more than one OAD within 3 months prior to screening;
* Use of Thiazolidinedione (TZD) within 6 months prior to screening;
* Use of insulin within 3 months prior to screening; Note: Short time use (≤10 days) of insulin due to acute illness or surgery (eg, infectious disease) is allowed.
* Any previous treatment with lixisenatide (eg, participation in a previous study with lixisenatide) or any other GLP-1 receptor agonist;
* Type 1 diabetes mellitus
* Women of childbearing potential with no effective contraceptive method;
* Pregnancy or lactation;
* Laboratory findings at the time of screening:

oAmylase and/or lipase >3 times the upper limit of the normal laboratory range (ULN);

* ALT >3 ULN;
* Calcitonin ≥20 pg/mL (5.9 pmol/L);
* Positive serum pregnancy test in women of childbearing potential;
* History of acute or chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease;
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (eg, multiple endocrine neoplasia syndromes);
* Allergic reaction to metacresol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety over 24 and 52 weeks assessed by treatment emergent adverse event (TEAE), vital signs, 12-lead electrocardiogram (ECG), and laboratory data. | from baseline to 24 weeks and 52 weeks

SECONDARY OUTCOMES:
Absolute change in HbA1c | from baseline to week 24 and week 52
Absolute change in fasting plasma glucose | from baseline to week 24 and week 52
Absolute change in body weight | from baseline to week 24 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- Japan (30):
  - Investigational Site Number 392006, Adachi-Ku
  - Investigational Site Number 392005, Chiba
  - Investigational Site Number 392010, Chiyoda-Ku
  - Investigational Site Number 392003, Chuoh-Ku
  - Investigational Site Number 392004, Chūōku
  - Investigational Site Number 392015, Chūōku
  - Investigational Site Number 392012, Ebina-Shi
  - Investigational Site Number 392024, Higashiosaka-Shi
  - Investigational Site Number 392023, Kashiwara-Shi
  - Investigational Site Number 392008, Kawagoe-Shi
  - Investigational Site Number 392009, Kisarazu-Shi
  - Investigational Site Number 392002, Koganeishi
  - Investigational Site Number 392007, Koriyama-Shi
  - Investigational Site Number 392011, Mitaka-Shi
  - Investigational Site Number 392025, Nagoya
  - Investigational Site Number 392026, Nagoya
  - Investigational Site Number 392013, Ogawa-Machi, Hikigun
  - Investigational Site Number 392014, Ohta-Ku
  - Investigational Site Number 392022, Okawa-Shi
  - Investigational Site Number 392021, Osaka
  - Investigational Site Number 392028, Osaka
  - Investigational Site Number 392029, Osaka
  - Investigational Site Number 392030, Sapporo
  - Investigational Site Number 392018, Sendai
  - Investigational Site Number 392001, Shinjuku-Ku
  - Investigational Site Number 392020, Suita-Shi
  - Investigational Site Number 392017, Toshima-Ku
  - Investigational Site Number 392027, Toyonaka-Shi
  - Investigational Site Number 392016, Yokohama
  - Investigational Site Number 392019, Yokohama